CLINICAL TRIAL: NCT03968757
Title: Assessing the Safety and Performance of the easyEndoTM Universal Linear Cutting Stapler in Laparoscopic Gastric Bypass Surgery: a Monocentric Post-market Observational Study
Brief Title: Assessing the Safety and Performance of the easyEndoTM Universal Linear Cutting Stapler in Laparoscopic Gastric Bypass Surgery
Status: Completed | Type: Observational
Sponsor: Duomed (Industry)
Responsible Party: Sponsor
Other Study IDs: STAP-D
Record Dates: First submitted 2019-05-22; First posted 2019-05-30 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Roux-en-Y Gastric Bypass; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Obese patients eligible for laparoscopic RYGB surgery.
  Interventions: Device: easyEndoTM Universal Linear Cutting Stapler and reloads (Ezisurg Medical)

INTERVENTIONS:
Device: easyEndoTM Universal Linear Cutting Stapler and reloads (Ezisurg Medical) — Device for creation of anastomoses during laparoscopic RYGB surgery manufactured by Ezisurg Medical.

SUMMARY:
The purpose of this observational registry is to evaluate the safety and performance of the easyEndoTM Universal Linear Cutting Stapler and reloads from Ezisurg Medical used in laparoscopic RYGB surgery to create anastomoses. The goal of the study will be achieved by assessing the device performance and reporting of peri- and postoperative complications in a prospectively maintained database.

ELIGIBILITY:
Inclusion Criteria:

1. Age at study entry is at least 18 years.
2. Patient must sign and date the informed consent form prior to the index-procedure. If the patient is not able to give informed consent, a legally authorized representative must give informed consent on his/her behalf.
3. Patient has a BMI ≥ 35 kg/m2 with one of more related co-morbidities.
4. Patient has a BMI ≥ 40 kg/m2.

Exclusion Criteria:

1. Patient is pregnant.
2. History of bariatric surgery.
3. Patient is known to be, or suspected of being unable to comply with the study protocol or proposed follow-up visits (e.g. no permanent address, known to be non-compliant or presenting an unstable psychiatric history).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese patients eligible for laparoscopic RYGB surgery. This registry will collect data from 150 laparoscopic RYGB procedures in which anastomoses are created with the easyEndoTM Universal Linear Cutting Stapler and reloads (Ezisurg Medical).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-07-04 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-06-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of the easyEndoTM Universal Linear Cutting Stapler and reloads (Ezisurg Medical) | at index-procedure
  Number of participants with peri-operative anastomotic leaks and intraluminal/intraperitoneal bleeding.
To evaluate the safety of the easyEndoTM Universal Linear Cutting Stapler and reloads (Ezisurg Medical) | at discharge, up to 1 week
  Number of participants with post-operative anastomotic leaks and intraluminal/intraperitoneal bleeding.
To evaluate the safety of the easyEndoTM Universal Linear Cutting Stapler and reloads (Ezisurg Medical) | at 6 weeks follow-up
  Number of participants with post-operative anastomotic leaks and intraluminal/intraperitoneal bleeding.
To evaluate the safety of the easyEndoTM Universal Linear Cutting Stapler and reloads (Ezisurg Medical) | at 6 months follow-up
  Number of participants with post-operative anastomotic leaks and intraluminal/intraperitoneal bleeding.
To evaluate the safety of the easyEndoTM Universal Linear Cutting Stapler and reloads (Ezisurg Medical) | at 12 months follow-up
  Number of participants with postoperative anastomotic leaks and intraluminal/intraperitoneal bleeding.
To evaluate the safety of the easyEndoTM Universal Linear Cutting Stapler and reloads (Ezisurg Medical) | at 24 months follow-up
  Number of participants with post-operative anastomotic leaks and intraluminal/intraperitoneal bleeding.

SECONDARY OUTCOMES:
To evaluate the performance of the easyEndoTM Universal Linear Cutting Stapler and reloads (Ezisurg Medical) | at index-procedure
  Number of procedures with technical success, defined as laparoscopic Roux-en-Y gastric bypass formation as intended without technical difficulties and without conversion to open laparotomy.
To evaluate the performance of the easyEndoTM Universal Linear Cutting | at index-procedure
  Assessment of device performance (e.g. sharpness of the blade, staple-line formation, etc.).
To evaluate the efficacy of the laparoscopic RYGB surgery | at index-procedure
  Number of participants with peri-operative complications such as but not limited to: peritonitis, anastomotic stenosis/stricture, internal hernia, small bowel obstruction, ulceration, fistula formation, ventral hernia, iatrogenic splenic injury, wound infection, pneumonia, pulmonary embolism, kidney failure, gallstones, arrhythmia, stroke, infarction, death.
To evaluate the efficacy of the laparoscopic RYGB surgery | at discharge, up to 1 week
  Number of participants with post-operative complications such as but not limited to: peritonitis, anastomotic stenosis/stricture, internal hernia, small bowel obstruction, ulceration, fistula formation, ventral hernia, iatrogenic splenic injury, wound infection, pneumonia, pulmonary embolism, kidney failure, gallstones, arrhythmia, stroke, infarction, death.
To evaluate the efficacy of the laparoscopic RYGB surgery | at 6 weeks follow-up
  Number of participants with post-operative complications such as but not limited to: peritonitis, anastomotic stenosis/stricture, internal hernia, small bowel obstruction, ulceration, fistula formation, ventral hernia, iatrogenic splenic injury, wound infection, pneumonia, pulmonary embolism, kidney failure, gallstones, arrhythmia, stroke, infarction, death.
To evaluate the efficacy of the laparoscopic RYGB surgery | at 6 months follow-up
  Number of participants with post-operative complications such as but not limited to: peritonitis, anastomotic stenosis/stricture, internal hernia, small bowel obstruction, ulceration, fistula formation, ventral hernia, iatrogenic splenic injury, wound infection, pneumonia, pulmonary embolism, kidney failure, gallstones, arrhythmia, stroke, infarction, death.
To evaluate the efficacy of the laparoscopic RYGB surgery | at 12 months follow-up
  Number of participants with post-operative complications such as but not limited to: peritonitis, anastomotic stenosis/stricture, internal hernia, small bowel obstruction, ulceration, fistula formation, ventral hernia, iatrogenic splenic injury, wound infection, pneumonia, pulmonary embolism, kidney failure, gallstones, arrhythmia, stroke, infarction, death.
To evaluate the efficacy of the laparoscopic RYGB surgery | at 24 months follow-up
  Number of participants with post-operative complications such as but not limited to: peritonitis, anastomotic stenosis/stricture, internal hernia, small bowel obstruction, ulceration, fistula formation, ventral hernia, iatrogenic splenic injury, wound infection, pneumonia, pulmonary embolism, kidney failure, gallstones, arrhythmia, stroke, infarction, death.
To evaluate the efficacy of the laparoscopic RYGB surgery | at discharge, up to 1 week
  Number of participants with bariatric surgery related re-interventions since the laparoscopic RYGB procedure.
To evaluate the efficacy of the laparoscopic RYGB surgery | at 6 weeks follow-up
  Number of participants with bariatric surgery related re-interventions since the laparoscopic RYGB procedure.
To evaluate the efficacy of the laparoscopic RYGB surgery | at 6 months follow-up
  Number of participants with bariatric surgery related re-interventions since the laparoscopic RYGB procedure.
To evaluate the efficacy of the laparoscopic RYGB surgery | at 12 months follow-up
  Number of participants with bariatric surgery related re-interventions since the laparoscopic RYGB procedure.
To evaluate the efficacy of the laparoscopic RYGB surgery | at 24 months follow-up
  Number of participants with bariatric surgery related re-interventions since the laparoscopic RYGB procedure.
To evaluate the efficacy of the laparoscopic RYGB surgery | at 6 weeks follow-up
  Change of patient's weight
To evaluate the efficacy of the laparoscopic RYGB surgery | at 6 months follow-up
  Change of patient's weight
To evaluate the efficacy of the laparoscopic RYGB surgery | at 12 months follow-up
  Change of patient's weight
To evaluate the efficacy of the laparoscopic RYGB surgery | at 24 months follow-up
  Change of patient's weight

CONTACTS AND LOCATIONS:
Locations (1):
- AZ Sint-Jan Brugge, Bruges, West Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No